CLINICAL TRIAL: NCT07259850
Title: Associations of Postoperative Delirium With Perioperative Frailty Worsening and Their Combined Effect on 1-Year Mortality in Older Surgical Patients: A Prospective Cohort Study
Brief Title: Associations of Postoperative Delirium With Perioperative Frailty Worsening and Their Combined Effect on 1-Year Mortality in Older Surgical Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yanhong Liu, Deputy Chief of administration, Anesthesiology, Chinese PLA General Hospital
Other Study IDs: PLAGH - FRAIL
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Delirium (POD); Frailty at Older Adults; Mortality; Recovery of Function
Keywords: postoperative delirium; frailty; older adults; one year mortality; frailty worsening
MeSH Terms: conditions — Emergence Delirium; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A retrospective cohort study based on prospectively collected data.: Patients were classified into POD and non-POD groups according to the occurrence of delirium within 7 days after surgery. The study examined the association between POD and worsened frailty at 1 month, and their combined effect on 1-year mortality.

SUMMARY:
Postoperative delirium (POD) is a frequent complication in older surgical patients and is associated with adverse outcomes, while frailty is also highly prevalent during the perioperative period. This study aimed to determine whether POD accelerates perioperative frailty worsening and to assess the effect of their coexistence on 1-year mortality.

ELIGIBILITY:
Inclusion criteria:

1. Aged ≥65 years;
2. Scheduled for elective non-cardiac, non-neurosurgical procedures;
3. Consented to undergo preoperative health and functional state assessments.

Exclusion criteria:

1. Had severe dementia, language disorders, significant hearing or visual impairments, or were in a coma;
2. Had Mini-Mental State Examination (MMSE) scores below the established educational thresholds: <18 for illiterate individuals, <21 for those with primary education (≤6 years), and <25 for those with secondary education or higher (>6 years)
3. Underwent local anesthesia or monitored anesthesia care;
4. Had an operative time ≤30 minutes;
5. Incomplete preoperative FRAIL scale assessment;
6. Missing postoperative delirium data;
7. Incomplete FRAIL scale assessment at 1 month postoperatively.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients were divided into postoperative delirium (POD) and non-POD groups based on delirium occurrence within 7 days after surgery. Follow-up assessments were conducted at 30 days and 1 year postoperatively to evaluate frailty change and survival outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 6196 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome was worsened frailty at one month after surgery. | At one month after surgery.
  Frailty was assessed preoperatively by trained researchers using the FRAIL scale, which includes five items: fatigue, resistance, ambulation, illnesses, and weight loss. Each item scores 0 or 1, for a total of 0-5 points, with higher scores indicating greater frailty. Patients were categorized as robust (0), pre-frail (1-2), or frail (3-5). A follow-up frailty assessment was conducted one month postoperatively via telephone. Frailty change was defined as the difference between postoperative and preoperative scores: ≤0 indicated stable/improved frailty, and >0 indicated worsened frailty.

SECONDARY OUTCOMES:
The secondary outcome was 1-year all-cause mortality. | At one year after surgery.
  A structured telephone follow-up was conducted one year after surgery to determine outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- 28 Fuxing Road, Haidian District, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No